CLINICAL TRIAL: NCT02708797
Title: Brainstem Grey Matter and Cerebral Autoregulation in Migraine With Aura : a MRI and Transcranial Doppler.
Brief Title: Brainstem Grey Matter and Cerebral Autoregulation in Migraine With Aura.
Acronym: MINOTAURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/15/7815; 2015-A01982-47 (Other: ID-RCB)
Record Dates: First submitted 2016-03-09; First posted 2016-03-15 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Migraine With Aura
Keywords: Cerebral autoregulation; MRI; VBM; Doppler Transcranial
MeSH Terms: conditions — Migraine with Aura | interventions — Magnetic Resonance Spectroscopy; Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Migraine with aura Patients (Other): Patients with migraine with aura will be studied 30 days after the pre inclusion visit with both magnetic resonance imaging and Transcranial Doppler.
  Interventions: Other: Magnetic resonance imaging; Other: Transcranial Doppler
- Controls (Other): Control group with healthy volunteers will be studied 30 days after the pre inclusion visit with both magnetic resonance imaging and Transcranial Doppler.
  Interventions: Other: Magnetic resonance imaging; Other: Transcranial Doppler

INTERVENTIONS:
Other: Magnetic resonance imaging — Patients and controls will first be studied with MRI. The total duration of MRI is about 60mn. These technic is not invasive.
Other: Transcranial Doppler — Patients and controls will first be studied with TCD. The total duration of TCD is about 60mn. These technic is not invasive.

SUMMARY:
Migraine with aura (MA) is an independent risk factor for stroke and is associated with silent brain infracts and T2 white matter hyperintensities on MRI. Previous studies using Transcranial Doppler (TCD) have shown an impairment of cerebral autoregulation in MA patients. Studies with positron emission tomography have demonstrated an activation of brain stem areas during migraine attack. An increased density of brain stem grey matter as measured on MRI with voxel based morphometry (VBM) has been found in MA patients. As brain arteries and arterioles are innervated by ascending tracts from aminergic brainstem nuclei, th study hypothesize a negative correlation between the density of brainstem nuclei and the efficiency of cerebral autoregulation in MA patients compared with controls.

Brainstem grey matter density will be studied with a MRI Philips 3 Tesla with a 32-channel antenna and voxel-based morphometry (VBM) cerebral autoregulation will be measured in the time domain using Transcranial Doppler (TCD) and the Mx method.

MA patients will be studied in a headache-free period. MRI and Transcranial Doppler (TCD) are non-invasive technics and will be performed on the same day.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with aura patients : fulfilling the International Classification of Headache Disorders-3 beta criteria of MA
* Control group : Gender- and age-matched subjects without history of migraine with or without aura or any other headache

Exclusion Criteria:

* History of illness or injury of central or peripherical nervous system
* Previous history of a disease potentially impairing cerebral autoregulation (diabetes, sleep apnea syndrome, uncontrolled hypertension, cardiac arrhythmia, hearth failure, carotid stenosis)
* Contraindications related to MRI
* Absence of temporal acoustic window
* Pregnancy

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Correlation between the density of the pontine grey matter evaluated with resonance magnetic imaging, and cerebral autoregulation measured with Transcranial Doppler in migraine with aura patients and controls. | 30 days after the pre-inclusion visit
  Resonance magnetic imaging use voxel base morphometry and Transcranial doppler use the coefficient mx calculation.

SECONDARY OUTCOMES:
Comparison of brainstem grey matter density between migraine with aura patients and controls with magnetic resonance imaging | 30 days after pre-inclusion visit
  Comparison will be done with software using voxel based morphometry (VBM) function in addition of imaging with resonance magnetic imaging.
Comparison of cerebral autoregulation between migraine with aura patients and controls with Transcranial Doppler | 30 days after pre-inclusion visit
  Comparison will be done using the calculation of mx coefficient in addition of imaging with Transcranial Doppler.
Comparison of cerebrovascular reactivity to carbon dioxide between migraine with aura patients and controls with Transcranial Doppler | 30 days after pre-inclusion visit
  Comparison will be done using voluntary apnea test in addition of imaging with Transcranial Doppler.
Comparison of morphological abnormalities between migraine with aura patients and controls with resonance magnetic imaging. | 30 days after pre-inclusion visit
  Comparison will be done using T2 white matter hyperintensities and silent brain infracts on resonance magnetic imaging.
Comparison of baroreflex sensitivity between migraine with aura patients and controls with Transcranial Doppler | 30 days after pre-inclusion visit
Association between grey matter density and morphological abnormalities on resonance magnetic imaging | 30 days after pre-inclusion visit
  Association will be determined using T2 white matter hyperintensities, silent brain infracts and voxel based morphometry function of software
Association between cerebral autoregulation and morphological abnormalities on magnetic resonance imaging | 30 days after pre-inclusion visit
  Association will be determined using T2 white matter hyperintensities, silent brain infracts and calculation of mx coefficient
Relation between baroreflex sensitivity and cerebral autoregulation with Transcranial Doppler. | 30 days after pre-inclusion visit
  Relation will be determined using the calculation of mx coefficient in addition of imaging with Transcranial Doppler

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LARRUE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gollion C, Nasr N, Fabre N, Barege M, Kermorgant M, Marquine L, Larrue V. Cerebral autoregulation in migraine with aura: A case control study. Cephalalgia. 2019 Apr;39(5):635-640. doi: 10.1177/0333102418806861. Epub 2018 Oct 8. PMID 30296840
- [Derived] Gollion C, Lerebours F, Nemmi F, Arribarat G, Bonneville F, Larrue V, Peran P. Insular functional connectivity in migraine with aura. J Headache Pain. 2022 Aug 19;23(1):106. doi: 10.1186/s10194-022-01473-1. PMID 35982396